CLINICAL TRIAL: NCT01716481
Title: Intravenous Administration of Autoserum-cultured Autologous Mesenchymal Stem Cells in Ischemic Stroke: A Single Center, Randomized, Open Label, Prospective, Phase 3 Study
Brief Title: The STem Cell Application Researches and Trials In NeuroloGy-2 (STARTING-2) Study
Acronym: STARTING-2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Pharmicell Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Oh Young Bang, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-10-047
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Stroke, Ischemic
Keywords: Stroke; Mesenchymal stem cells; Stem cells; Neurogenesis
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cell treatment (Experimental)
  Interventions: Other: Mesenchymal stem cell
- Standard treatment (No Intervention)

INTERVENTIONS:
Other: Mesenchymal stem cell — intravenous transplantation of autologous mesenchymal stem cells expanded with autologous serum
  Arms: Mesenchymal stem cell treatment

SUMMARY:
The objectives of this study was to test hypothesis that ischemic stroke patients having moderate to severe persistent neurologic deficit will have better outcomes with intravenous transplantation of autologous mesenchymal stem cells (MSCs) expanded with autologous serum that is obtained at acute phase of stroke than patients receiving standard treatment.

DETAILED DESCRIPTION:
In this study, we will use autologous 'ischemic' serum that obtained at the earliest time point as possible (immediate after randomization) for the purpose of ischemic preconditioning. We have recently conducted preclinical studies on the effects of ischemic preconditioning on the MSC functions. We have evaluated the characteristics of rat MSCs after culture with fetal bovine serum (FBS) or serum obtained from rat stroke model. Compared to FBS, the use of serum obtained from rat stroke model resulted in more rapid expansion of MSCs, which reduces cell preparation time by increase in G2/M phase, decreased cell death/senescence, increased trophic factor secretion, and increased migration capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women (women must be of non-child bearing potential), age 30-75 yrs.
2. Have a stroke that is observed within 90 days of the onset of symptoms
3. Radiologically

   1. Relevant lesions within the middle cerebral artery territory (MCA) as assessed using diffusion-weighted imaging (DWI).
   2. The maximum diameter of the stroke region in any dimension must be ≥15 mm.
   3. Not involving more than a half of the ipsilateral periventricular zone
4. Clinically (National Institutes of Health stroke scale, NIHSS)

   1. Moderate-to severe persistent neurologic deficit (NIHSS of 6-21 inclusive)
   2. New onset of extremity paresis on the affected side, defined as a score of 2-4 on the NIHSS Motor Arm (item 5) or Leg (item 6) question.
   3. Must be alert or drowsy but easily arousable as defined by score of 0-1 on the NIHSS Level of Consciousness question (item 1).
   4. "Slow recovery" defined as Change in NIHSS ≤1 point/3 days
5. Willingness

   1. Reasonable likelihood of receiving standard physical, occupational and speech rehabilitation therapy as indicated for the post stroke deficits.
   2. Able to participate in the evaluation process to the point of accurate assessment.
   3. Willing and able to comply with scheduled visits, lifestyle guidelines, treatment plan, laboratory tests, and other study procedures.
   4. Evidence of a personally signed and dated informed consent document.

Exclusion Criteria:

1. Presence of significant disability prior to the current stroke. Significant disability is defined as having a pre-stroke modified Rankin score of 2 or more.
2. Have a stroke that is either

   1. lacunar infarction
   2. Hematologic cause of stroke
   3. Recurrent or progressive stroke within 1 week at the time of screening.
3. Hematologic disorders or bone marrow suppression.
4. Have a severe medical illness

   1. Severe heart failure
   2. Severe febrile illness
   3. Hepatic or renal dysfunction
   4. Active cancer
   5. Any evidence of chronic co-morbid condition or unstable acute systemic illnesses which, in the opinion of the investigator, could shorten the subject's survival or limit ability to complete the study.
5. Presence of human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), or syphilis on admission blood tests
6. Presence of depression that is active and not adequately controlled such that it interfere with major activities of daily living immediately prior to the current stroke.
7. Presence of dementia prior to the current stroke that is likely to confound clinical evaluation.
8. Pregnant females as determined by positive urine human chorionic gonadotropin (hCG) test or lactating females.
9. Subjects considered unwilling or unable to comply with the procedures and study visit schedule outlined in the protocol
10. Subjects unwilling to undergo bone marrow aspiration

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Categorical shift in modified Rankin scale (mRS) | 90 days after the cell treatment
  Categorical shift in mRS at 90 days after the cell treatment

SECONDARY OUTCOMES:
Change of National Institutes of Health stroke scale (NIHSS) | 90 days after the cell treatment
  Change of NIHSS between pre- and post-treatment 90 days
Early improvement of National Institutes of Health stroke scale (NIHSS) | 14 days after the cell treatment
  ≥5 points improvement or score of 0-2 on NIHSS score at 14 days after treatment
Dichotomized modified Rankin scale (mRS) | 90 days after the cell treatment
  mRS ≤2 at 90 days after treatment
Change of modified Rankin scale (mRS) | 90 days after the cell treatment
  Change of mRS between pre- and post-treatment 90 days
Dichotomized modified Barthel index (mBI) | 90 days after the cell treatment
  mBI ≥60 at 90 days after treatment
Change of modified Barthel index (mBI) | 90 days after the cell treatment
  Change of mBI between pre- and post-treatment 90 days
Change of gross motor function | 90 days after the cell treatment
  Change of Gross motor function (Motricity index and Fugl-Meyer assessment)between pre- and post-treatment 90 days
Change of Fine motor function | 90 days after the cell treatment
  Change of Fine motor function (Purdue Pegboard test and Box and block test) between pre- and post-treatment 90 days
Change of Mobility | 90 days after the cell treatment
  Change of Mobility (Functional ambulatory category and 10m-Gait speed) between pre- and post-treatment 90 days
Change of mini-mental status exam (MMSE) | 90 days after the cell treatment
  Change of MMSE between pre- and post-treatment 90 days
Change of quality of life | 90 days after the cell treatment
  Change of EuroQol 5d (EQ-5D) between pre- and post-treatment 90 days
Safety outcome | During 90 days after the cell treatment
  1. Death: All causes of death
  2. Recurrence: Recurrent stroke or transient ischemic attack
  3. The immediate reaction:
     Allergic reactions (tachycardia, fever, skin eruption, leukocytosis) Local complications (hematoma or local infection at the site of bone marrow aspiration) Vascular obstruction (tachypnea, oliguria, or peripheral vascular insufficiency) Systemic complications (infections,laboratory findings).
  4. Long-term adverse effects possibly related to MSC treatment Tumor formation (physical examination, plain x-ray, f/u MRI at 90 days after treatment), Aberrant connections (newly diagnosed seizure or arrhythmia)

OTHER OUTCOMES:
Exploration of biomarkers | During 90 days after the cell treatment
  SDF(stromal cell-derived factor)-1ɑ (chemokine) S100ß (protection and regeneration) HIF(Hypoxia-inducible factor)-1 (preconditioning) Circulating MSCs and MSC-derived microparticles (CD105-CXCR4(C-X-C chemokine receptor type 4)-PS(phosphoserine)) BDNF (Brain-derived neurotrophic factor) levels and it's polymorphism, and VEGF (Vascular endothelial growth factor) levels
  Resting-state functional MRI & Diffusion tensor imaging

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Bang OY, Kim EH, Cho YH, Oh MJ, Chung JW, Chang WH, Kim YH, Yang SW, Chopp M. Circulating Extracellular Vesicles in Stroke Patients Treated With Mesenchymal Stem Cells: A Biomarker Analysis of a Randomized Trial. Stroke. 2022 Jul;53(7):2276-2286. doi: 10.1161/STROKEAHA.121.036545. Epub 2022 Mar 28. PMID 35341320
- [Derived] Lee J, Chang WH, Chung JW, Kim SJ, Kim SK, Lee JS, Sohn SI, Kim YH, Bang OY; STARTING-2 Collaborators. Efficacy of Intravenous Mesenchymal Stem Cells for Motor Recovery After Ischemic Stroke: A Neuroimaging Study. Stroke. 2022 Jan;53(1):20-28. doi: 10.1161/STROKEAHA.121.034505. Epub 2021 Sep 29. PMID 34583525
- [Derived] Chung JW, Chang WH, Bang OY, Moon GJ, Kim SJ, Kim SK, Lee JS, Sohn SI, Kim YH; STARTING-2 Collaborators. Efficacy and Safety of Intravenous Mesenchymal Stem Cells for Ischemic Stroke. Neurology. 2021 Feb 16;96(7):e1012-e1023. doi: 10.1212/WNL.0000000000011440. Epub 2021 Jan 20. PMID 33472925
- [Derived] Kim SJ, Moon GJ, Chang WH, Kim YH, Bang OY; STARTING-2 (STem cell Application Researches and Trials In NeuroloGy-2) collaborators. Intravenous transplantation of mesenchymal stem cells preconditioned with early phase stroke serum: current evidence and study protocol for a randomized trial. Trials. 2013 Oct 1;14:317. doi: 10.1186/1745-6215-14-317. PMID 24083670